CLINICAL TRIAL: NCT04065568
Title: An Interactive Distance Solution for Stroke Rehabilitation in the Home Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The pandemic. Collected data will presented as a pilot RCT.
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DISKO/STRADA
Record Dates: First submitted 2019-04-09; First posted 2019-08-22 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Stroke Rehabilitation
Keywords: Stroke; Rehabilitation; Medical technology
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A randomized controlled intervention study.
Who Masked: Outcomes Assessor
Masking Description: Baseline and outcome will be assessed by blinded physiotherapists not involved in the intervention, who will be trained to be synchronized in the assessment procedures and to follow the same standardised protocol to assure consistency both at the Danderyd Hospital and Stockholm Sjukhem site.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The patient will receive conventional out patient rehabilitation after discharge to the home after stroke. In addition an individualized training program with gamified excercises for motor function will be set and followed up by clincians using video communication, as part of the DISKO-tool. Patients are instructed to train self sufficiently 5 days a week and will be supervised by the treating physiotherapist. The intervention will last for 6 weeks.
  Interventions: Device: DISKO-tool
- Control group (No Intervention): Conventional rehabilitation in primary care after discharge to the home after stroke.

INTERVENTIONS:
Device: DISKO-tool — The training program will be based on the initial assessments of functioning and disability and the patients' performance of the test exercises. Type and number of exercises per session, level of difficulty and number of repetitions (including proportion of repetitions to the right and left side of the body) will be set. The set training program is thereafter introduced and evaluated during the first follow-up by video communication with the patients.
  Arms: Intervention group

SUMMARY:
Equal access to evidence based rehabilitation in the stroke population is a challenge. Home based solutions including telerehabilitation is a promising strategy to meet these needs. However, the tools must be customized for persons with stroke and the technologies developed to serve rehabilitation purposes. The DISKO-tool was developed to enable efficient, continuous training in the home setting with health professional follow ups of training and training results after stroke via video link. The tool has in a preliminary study proved feasible and safe in different phases after stroke. The functional effect of using the DISKO-tool added to conventional rehabilitation in the home setting is yet to be explored. Thus, the aim of this study is to explore the added value of using the DISKO-tool during rehabilitation in the home setting.

DETAILED DESCRIPTION:
Aim:The DISKO-tool was developed to enable efficient, continuous training in the home setting with health professional follow ups of training and training results after stroke via video link. The tool has in a preliminary study proved feasible and safe in different phases after stroke. The functional effect of using the DISKO-tool added to conventional rehabilitation in the home setting is yet to be explored. Thus, the aim of this study is to explore the added value of using the DISKO-tool during rehabilitation in the home setting.

Hypothesis to be tested: Participants who perform 6 weeks of intensive training supported by the DISKO-tool in addition to the regular stroke rehabilitation interventions, gain a higher level of functioning compared to the control group with regular rehabilitation interventions.

Study design: A randomized controlled intervention study.

Participants and methods: 100 participants will be included in the study 3-6 months after stroke and after informed consent. The participants are recruited from primary care i.e. neuroteam and out-patient rehabilitation in Stockholm, Sweden. The included patients will be randomized to either 1) the intervention group (n=50) or 2) the control group (n=50). Based on previously published results on the BESTtest [14], a significance level of 5% and a power of 80%, 41 patients/treatment arm need to be included. With an expected minimal loss of participants per treatment arm, the study will require 50 patients/treatment arm.

After the baseline assessment, the patients will receive a first introduction to the DISKO-tool. Thereafter the DISKO-tool system is set up at the patients' home by the physiotherapist. For safety reasons, space requirements and convenience of the patients, the physiotherapist in dialogue with the patients will select the placement of the screen. During the home visit, the patients will receive a manual and are instructed and guided in how to use the DISKO-tool including turning on the screen, controlling the user interface and performing test exercises. Dates and times for follow-ups by video communication with the physiotherapist are scheduled. After the installation, the physiotherapist will design an individualized training program for each of the patients. The training program will be based on the initial assessments of functioning and disability and the patients' performance of the test exercises. Type and number of exercises per session, level of difficulty and number of repetitions (including proportion of repetitions to the right and left side of the body) will be set. The set training program is thereafter introduced and evaluated during the first follow-up by video communication with the patients. In both groups, patients are instructed to train self-sufficiently 5 days a week and will be supervised by the treating physiotherapist. The intervention will last for 6 weeks. The baseline and final testing will both be performed at the rehabilitation clinics.

The follow-ups, by video communication, will be registered by the physiotherapists in standardised logbooks. Data on conventional interventions will be retrieved from medical records. From the DISKO-tool, data regarding number of performed self-training sessions will be retrieved.

After the intervention, the physiotherapist's (also after informed consent) and patient's experience and perception of using the DISKO-tool will be assessed in a study specific questionnaire based on the results of the semi-structured interviews performed in the feasibility study that preceded this study.

ELIGIBILITY:
Inclusion Criteria:

* impaired motor function after stroke limiting activities of daily living but can walk indoors with or without supervision (functional ambulation category[ >FAC 3), can stand without support >2 min and are able to perform a forward reach of >12 cm in standing position,
* referred to a neuroteam for rehabilitation interventions in the home setting and/or out- patient rehabilitation at Stockholms sjukhem or Rehab Nordost Täby
* motivated to perform exercises in the home setting with the DISKO-tool and with recurrent supervision by a physiotherapist through video communication.

Exclusion Criteria:

* cognitive and/or speech impairment, limiting the ability to follow verbal and written training instruction or study information
* other disabling neurological disorder or other diagnosis prohibiting physical activity necessary when utilizing the DISKO tool
* impaired vision preventing orientation and reading instructions on a screen
* sufficient internet access in the home to participate in the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
BESTest -to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses balance

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses stroke-related neurologic impairments (0p no detected impairment, summed up to 34p max impairment)
Montreal Cognitive Assessment- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses mental function (0p max impairment summed up to 30p no detected impairment)
Modified Ashworth Scale- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses spasticity on a 6 point scale/muscle (0p no impairment, 5p max impairment/muscle)
Fugle-Meyr for lower and upper extremity- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses sensory and movement related functions in lower and upper extremity (0p max impairment summed up to 86p max no detected impairment (lower extremity) 126p max no detected impairment (upper extremity)
Functional Ambulation Category- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses independence in walking 0p nonfunctional, 5p independent Total score 0-5p
6 minutes walk test combined with the RPE-scale- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses walking endurance in meters walked
Timed Up and Go Test- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses gait and mobility (timed sek)
Falls Efficacy Scale- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses self perceived balance in every day life activities rated on an 11 point scale (0p not safe at all 10p completely safe). Total score: 0- 130 p
Barthel Index- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses independence in mobility and personal care (0p dependent 10/15p independent) Total score 0-100p
Stroke Impact Scale- to assess change | T1 (baseline, before start of intervention) T2 (after completion of the 6 week intervention) and T3 (6 months after completion of the intervention)
  Assesses self perceived impact of stroke on functioning and disability (domains: strength, hand function, ADL/IADL, Mobility, Commnication, Emotion, Memory/thinking, Participation rated on a 5 point scale (1p maximum impairment/limitation/restriction, 5p minimum impairment/limitation/restriction) Total score 0-100 p/domain calculated using an algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Palmcrantz, PhD, Study Director — Danderyd Hosptial; Jorgen Borg, Prof, Study Director — Danderyd Hospital; Elisabet Akesson, Assoc Prof, Study Director — Karolinska Institutet; Erika Franzén, Assoc Prof, Study Director — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm County
  - Stockholms sjukhem, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehn M, Hansson P, Sjolinder M, Boman IL, Folke M, Sommerfeld D, Borg J, Palmcrantz S. Users perspectives on interactive distance technology enabling home-based motor training for stroke patients. Stud Health Technol Inform. 2015;211:145-52. PMID 25980861
- [Result] Palmcrantz S, Borg J, Sommerfeld D, Plantin J, Wall A, Ehn M, Sjolinder M, Boman IL. An interactive distance solution for stroke rehabilitation in the home setting - A feasibility study. Inform Health Soc Care. 2017 Sep;42(3):303-320. doi: 10.1080/17538157.2016.1253015. Epub 2016 Dec 5. PMID 27918220